CLINICAL TRIAL: NCT04561778
Title: HIS-Purkinje Conduction System Pacing Optimized Trial of Cardiac Resynchronization Therapy
Acronym: HOT-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pugazhendhi Vijayaraman (Other)
Responsible Party: Sponsor-Investigator, Pugazhendhi Vijayaraman, Sponsor-Investigator, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-0831
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure，Congestive; Cardiomyopathies; Left Ventricular Dysfunction
Keywords: Heart Failure; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Ventricular Dysfunction, Left | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded to treatment arm. Echocardiographic evaluation will be performed by study physician blinded to lead placement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HOT-CRT (Active Comparator): Subjects randomized to HOT-CRT will undergo CRT as described below. His bundle pacing lead will be placed initially to achieve CRT. If complete resynchronization is achieved (BBB normalization) but capture thresholds are high (1.5-2V), the lead may be placed in the distal conduction system (left bundle branch area). If only partial QRS narrowing is achieved, a coronary sinus lead may be placed and LV timing may be optimized to achieve maximal resynchronization. This will be at the discretion of the implanting physician. Only FDA approved leads and devices will be used.
  Interventions: Device: HOT-CRT
- Biventricular Pacing (Active Comparator): Subjects randomized to biventricular pacing will undergo left ventricular lead placement in the coronary sinus venous branches.Only FDA approved leads and devices will be used.
  Interventions: Device: Biventricular Pacing

INTERVENTIONS:
Device: HOT-CRT — Subjects enrolled in the study will receive a permanent cardiac implantable electronic device (CIED) (CRT-pacemaker or CRT-defibrillator) as clinically indicated. Subjects randomized to HOT-CRT will have His bundle pacing lead placed initially to achieve CRT. If complete resynchronization is achieved (BBB normalization) but capture thresholds are high (1.5-2V), the lead may be placed in the distal conduction system (left bundle branch area). If only partial QRS narrowing is achieved, a coronary sinus lead may be placed and left ventricular timing may be optimized to achieve maximal resynchronization.
  Arms: HOT-CRT
Device: Biventricular Pacing — Subjects enrolled in the study will receive a permanent CIED (CRT-pacemaker or CRT-defibrillator) as clinically indicated. Subjects randomized to Biventricular pacing will undergo left ventricular lead placement in the coronary sinus venous branches.
  Arms: Biventricular Pacing

SUMMARY:
This is a randomized, prospective, single-blinded trial to determine the overall rate of successful His-Purkinje conduction system pacing Optimized Trial of Cardiac Resynchronization Therapy (HOT-CRT) versus biventricular pacing using coronary sinus lead (BVP) to compare acute and mid-term outcomes. Acute outcomes include change in QRS duration pre-and post-pacing (degree of QRS narrowing) and incidence of major periprocedural complications (pericardial tamponade, need for lead revision, etc.). Mid-term outcomes include echocardiographic response at 6 months along with a composite clinical outcome of heart failure hospitalization, ventricular arrhythmias, crossover, and all-cause mortality.

DETAILED DESCRIPTION:
This is a single-blinded study of 100 patients randomized to a strategy of His-Purkinje conduction system pacing Optimized Trial of Cardiac Resynchronization Therapy (HOT-CRT) versus biventricular pacing using coronary sinus (CS) lead (BVP). Both treatment options use standard-of-care, FDA-approved devices. The distinction is only in the allocation toward HOT-CRT and BVP. Treating physicians will be aware of assignment in order to facilitate routine device follow-up. Echocardiographic and electrocardiographic evaluation will also be performed in a blinded manner.

Cross-over is permitted between treatment group allocation if:

CS lead cannot be placed due to difficult cannulation of the CS, limited branches at the posterolateral or lateral wall, or phrenic nerve capture. These subjects may then cross-over to HOT-CRT.

HOT-CRT subjects may cross-over if His or left bundle pacing lead cannot be positioned with adequate stability and reasonable pacing output, or if optimal QRS narrowing cannot be achieved.

Implant procedure will be per routine percutaneous access, as is standard for pacemaker and Implantable Cardioverter Defibrillators (ICDs). . All subjects will receive an FDA-approved cardiac resynchronization therapy pacemaker or defibrillator device, as per standard of care outlined for the subject.

Follow-up will be performed at 2 weeks post-implant for incision check and device interrogation as is standard of care. In addition, routine device and clinical follow-up will be scheduled at 3 and 6 months. Electrocardiography (ECG) will be performed pre-implant, prior to hospital discharge, at 3 months, and 6 months. Echocardiography will be performed pre-implant and 6 months to evaluate for change in Left Ventricular Ejection Fraction (LVEF), chamber dimensions, volumes, and change in Left Ventricular (LV) end systolic volume index as is standard of care in the treatment of patients with advanced heart failure. New York Heart Association (NYHA) functional class and quality of life (utilizing the Kansas City Cardiomyopathy Questionnaire (KCCQ) and EQ 5D) will be assessed pre-implant and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Diagnosis is NYHA Class II, III, and ambulatory Class IV heart failure with either ischemic or nonischemic cardiomyopathy and patients with NYHA Class I symptoms and ischemic cardiomyopathy, with at least one of the following:

  * LV systolic dysfunction with LVEF ≤ 35% and Evidence of bundle branch block with QRS duration > 120 msec
  * LV systolic dysfunction with LVEF ≤ 50% and with need for >40% Right Ventricular (RV) pacing

Exclusion Criteria:

* Existing CRT device
* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Pregnancy
* Participation in other device trials
* Inability to complete study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pugazhendhi Vijayaraman, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vijayaraman P, Pokharel P, Subzposh FA, Oren JW, Storm RH, Batul SA, Beer DA, Hughes G, Leri G, Manganiello M, Jastremsky JL, Mroczka K, Johns AM, Mascarenhas V. His-Purkinje Conduction System Pacing Optimized Trial of Cardiac Resynchronization Therapy vs Biventricular Pacing: HOT-CRT Clinical Trial. JACC Clin Electrophysiol. 2023 Dec;9(12):2628-2638. doi: 10.1016/j.jacep.2023.08.003. Epub 2023 Sep 13. PMID 37715742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from Geisinger Wyoming Valley, Geisinger Medical Center, and Geisinger Community Medical Center. Investigators will identify eligible subjects, describe the study procedures and invite them to participate in the study. Informed Consent (ICF) will be provided to the subject and they will have ample time and opportunity to review and consider participation. Prior to performing any study procedures, the subject will sign the ICF and be considered enrolled at that point.
Pre-assignment Details: Subjects were screened to meet inclusion/exclusion criteria pre consent and post consent, pre implant. In some cases, a repeat echo was scheduled to obtain ejection fraction (EF) measurement as part of inclusion/exclusion criteria, and result was pending at time of consent, therefore when resulted and patient no longer met inclusion criteria, they were screen failed.
Groups:
- BiV Pacing: Patients randomized to biventricular pacing will undergo left ventricular lead placement in the coronary sinus venous branches
- HOT-CRT: Patients randomized to HOT-CRT will undergo CRT as described below. His bundle pacing lead will be placed initially to achieve CRT. If complete resynchronization is achieved (BBB normalization) but capture thresholds are high (1.5-2V), the lead may be placed in the distal conduction system (left bundle branch area). If only partial QRS narrowing is achieved, a coronary sinus lead may be placed and left ventricular (LV) timing may be optimized to achieve maximal resynchronization. This will be at the discretion of the implanting physician.
Period: Overall Study
Arm/Group | BiV Pacing | HOT-CRT
Started (originally 50 patients were randomized to each group, however according to the protocol, participants in the BiV Pacing arm may have crossed over to the HOT-CRT arm because BiV Pacing could not be achieved. * 50 patients randomized to BiV - 43 received BiV treatment * 50 patients randomized to HOTCRT - 57 received HOTCRT treatment * There were 11 cross overs in total, 9 from BiV to HOTCRT and 2 from HOTCRT to BiV) | 50 | 50
Cross Over to HOTCRT | 9 | 0
Cross Over to BiV | 0 | 2
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 50 patients randomized to BiV - 43 received BiV treatment 50 patients randomized to HOTCRT - 57 received HOTCRT treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | HOT-CRT | Biventricular Pacing | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years]
  All patients | 71 (13.4) | 68.9 (11.5) | 70 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  All patients: Female | 11 | 20 | 31
  All patients: Male | 39 | 30 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 42 | 38 | 80
Diabetes [Count of Participants; unit: Participants] | 26 | 23 | 49
Coronary Artery Disease [Count of Participants; unit: Participants] | 23 | 22 | 45
Atrial fibrillation [Count of Participants; unit: Participants] | 12 | 22 | 34
Chronic kidney disease [Count of Participants; unit: Participants] | 17 | 18 | 35
Nonischemic cardiomyopathy [Count of Participants; unit: Participants] | 30 | 31 | 61
Left bundle branch block [Count of Participants; unit: Participants] | 31 | 31 | 62
Left ventricular ejection fraction [Mean (Standard Deviation); unit: percent ejection fraction] | 30.1 (9.1) | 30.7 (9.3) | 30.4 (9.1)
QRS [Mean (Standard Deviation); unit: ms] | 164 (26) | 166 (28) | 165.0 (26.5)
New York Heart Association (NYHA) functional class [Mean (Standard Deviation); unit: units on a scale] — New York Heart Association functional class Range: I-IV I-No limitation of physical activity. II-Slight limitation of physical activity III-Marked limitation of physical activity IV-Symptoms of heart failure at rest. Any physical activity causes further discomfort Higher value represents worse clinical condition
  units on a scale | 2.5 (0.7) | 2.5 (0.7) | 2.5 (0.7)
Medications [Count of Participants; unit: Participants]
  Beta blocker | 45 | 47 | 92
  Aldosterone antagonist | 14 | 15 | 29
  Amiodarone | 9 | 8 | 17
  ACE | 22 | 13 | 35
  ARB | 10 | 5 | 15
  ARNI | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint
Description: Improvement in left ventricular ejection fraction (LVEF) - change in LVEF% measured by 2D echo at 6 months compared to baseline
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | HOT-CRT | Biventricular Pacing
Number analyzed (Participants) | 50 | 50
percent ejection fraction | 12.4 (7.3) | 8.0 (10.1)

2. Primary Outcome: Primary Safety
Description: Freedom from major complications or need for CRT lead revision - complication such as lead dislodgment, pericardial tamponade, pneumothorax, systemic embolism, phrenic nerve stimulation not correctable by programming
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HOT-CRT | Biventricular Pacing
Number analyzed (Participants) | 50 | 50
Participants | 49 | 48

3. Secondary Outcome: Secondary Composite
Description: Crossover, ventricular tachycardia (VT)/ventricular fibrillation (VF), Heart failure hospitalization (HFH) or death
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HOT-CRT | Biventricular Pacing
Number analyzed (Participants) | 50 | 50
Participants | 9 | 14

4. Secondary Outcome: Echocardiographic Response
Description: change in LVEF >5%
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HOT-CRT | Biventricular Pacing
Number analyzed (Participants) | 50 | 50
Participants | 35 | 27

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were monitored through the patient's study participation (about 6 months) and throughout the course of the study.
Description: An AE includes, but is not limited to, the following: Any clinically significant worsening of a preexisting condition. An AE occurring from abuse (e.g., use for nonclinical reasons) of a test article. An AE that has been associated with the discontinuation of the use of a test article.
  50 patients randomized to BiV - 43 received BiV treatment 50 patients randomized to HOTCRT - 57 received HOTCRT treatment
Arm/Group | HOT-CRT | Biventricular Pacing
All-Cause Mortality (participants affected / at risk) | 2/57 | 2/43
Serious Adverse Events (participants affected / at risk) | 17/57 | 32/43
Other Adverse Events (participants affected / at risk) | 0/57 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HOT-CRT (N=57) | Biventricular Pacing (N=43)
Threshold increase >1 V (Cardiac disorders) | 2 | 4
Lead dislodgement (Cardiac disorders) | 3 | 2
Stroke (Cardiac disorders) | 0 | 0
Infection (Infections and infestations) | 0 | 1
Late perforation into left ventricle (Cardiac disorders) | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0
Phrenic nerve stimulation (Cardiac disorders) | 0 | 4
Hematoma requiring evacuation (Surgical and medical procedures) | 0 | 1
Secondary composite clinical endpoint (Cardiac disorders) | 9/50 | 14 — Heart failure hospitalization, treatment crossover, VT/VF requiring implantable cardioverter-defibrillator (ICD) therapy
Total (Cardiac disorders) | 3 | 10

LIMITATIONS AND CAVEATS:
This was a small randomized pilot clinical trial performed in a single health system experienced in HOTCRT. This study was limited to 6 months of follow-up care and was not powered to detect differences in clinical outcomes. The study population was not diverse and included only a small number of women. Future large multicenter randomized controlled studies with longer follow-up times are needed for a comparison of long-term clinical outcomes between HOTCRT and BiV pacing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT04561778/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04561778/ICF_001.pdf